CLINICAL TRIAL: NCT05560932
Title: HIV and Alcohol Research Center Focused on Polypharmacy (HARP) Pilot 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Justice 090622; P01AA029545-03 (NIH); P01 AA029545-03 sub 9238 (Other Grant/Funding Number: Sub Award P01 AA029545-03)
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: HIV; Alcohol Use
MeSH Terms: conditions — Alcohol Drinking | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIV Medications and Alcohol Use (Experimental): Participants with HIV who take 5 or more medications and currently (within the past month) consume alcohol
  Interventions: Behavioral: IMB-motivational interviewing (MI) techniques (IMB-MI)

INTERVENTIONS:
Behavioral: IMB-motivational interviewing (MI) techniques (IMB-MI) — The clinical pharmacist will employ MI in informational, participant-centered discussions in which the clinical pharmacist and participant collaboratively discuss the harms of drinking and polypharmacy (specifically alcohol interactive medications), symptoms associated with alcohol and specific medications, and how to mitigate these harms. Motivational elements include messages highlighting the participant's personal risk of bothersome symptoms from their use of alcohol and level of polypharmacy, attitude change elements to improve attitudes toward the intended behavior change, social normative support for the intended behavior change including identification of people who can support the participant in this process, and a menu of options for referrals for skill building (e.g. Social Work, meeting with the clinical pharmacist at their clinic, follow-up with the HIV clinician, alcohol-reduction programs, based on what is locally available as part of VA-based care).

SUMMARY:
This pilot intervention will consist of a brief intervention for patients with HIV who take 5 or more medications and currently (within the past month) consume alcohol. The focus of this pilot will be on bothersome symptoms and the impact of alcohol use and medications on these symptoms. The rationale is that any alcohol use may interact with medications in serious ways leading to adverse outcomes, including bothersome symptoms.

DETAILED DESCRIPTION:
Additional outcomes were added at results entry.

ELIGIBILITY:
Inclusion Criteria:

* participants in both Veterans Aging Cohort Study (VACS) and Medications, Alcohol, and Substance use in HIV (MASH) studies
* prescribed 5 or more medications AND who either have a positive PEth value (8+) or a self-reported AUDIT-C value consistent with current alcohol use (score >0)

Exclusion Criteria:

* Alcohol use disorder (AUD) diagnosis in the past 12 months or who test positive for AUD on the Alcohol Symptom Checklist for moderate or severe AUD (score of 4 or more)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Justice, MD, PhD, Principal Investigator — Yale University
Locations (1):
- West Haven CT Veterans Administration, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
The data will not be shared by placing it in a data repository, but will be shared with those who submit a reasonable request .

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 enrolled, 12 did not complete any study activities, 38 started and received intervention
Period: Overall Study
Arm/Group | HIV Medications and Alcohol Use
Started | 38 (received intervention)
Intervention Only | 3 (completed intervention but did not complete post-intervention assessments)
Completed | 35 (completed study per protocol)
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 33
  White | 3
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 38
Education [Count of Participants; unit: Participants]
  High School Graduate | 14
  Some College | 13
  College Graduate | 11

OUTCOME MEASURES:

1. Primary Outcome: Enrollment to Assess Feasibility
Description: Number of participants that enrolled and provided informed consent
Time Frame: baseline
Population: 50 participants were enrolled. 12 did not complete any study activities.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 50
Participants | 50

2. Primary Outcome: Completion to Assess Feasibility
Description: Number of participants that completed the full pilot intervention
Time Frame: Study completion (Post-intervention Day 30)
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 38
Participants | 35

3. Primary Outcome: Qualitative Interviews to Assess Feasibility
Description: Number of participants that successfully completed the qualitative interviews
Time Frame: Study completion (within one to four weeks after Post-intervention Day 30)
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 38
Participants | 20

4. Primary Outcome: Change in Bothersome Symptoms From Baseline Using the HIV Symptoms Index
Description: The HIV Symptoms Index is a 20-item, self-reported measure that assesses presence and perceived distress linked to symptoms associated with HIV or HIV treatment. There are 5 possible responses: 0 = I don't have this symptom; 1 = It doesn't bother me; 2 = It bothers me a little; 3 = It bothers me; and 4 = It bothers me a lot, for each HIV symptom. Presented here is the number of bothersome symptoms with improvement on post-intervention Day 1 and post-intervention Day 30.
Time Frame: baseline, post-intervention Day 1, Post-intervention Day 30
Measure: Number; unit: symptoms
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 35
symptoms
  Symptoms with improvement from baseline to post intervention Day 1. | 1
  Symptoms with improvement from baseline to post-intervention Day 30. | 5

5. Primary Outcome: Number of Participants That Completed Both PEth Tests to Assess Acceptability.
Description: Change in alcohol levels assessed measuring PEth levels in the blood. PEth testing uses blood to measure alcohol use by detecting direct alcohol biomarkers in the bloodstream. A positive test indicates alcohol use.
Time Frame: baseline and Post-intervention Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 38
Participants | 35

6. Primary Outcome: Participants Readiness to Change Prescribed Medications
Description: The mean score of participants responses by self report. Participants were asked "If your provider felt it was a good idea, how ready are you to decrease your medications?", "If your provider felt it was a good idea, how important is it for you to decrease your medications?", and "If your provider felt it was a good idea, how confident are you that you can decrease your medications?" Each question is scored on a 1-10 scale (1=not at all ready, 10=extremely ready). Total score range for each question is 1-10 with higher scores indicating better outcomes.
Time Frame: baseline, immediately post intervention (day 1) and Post-intervention Day 30
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 38
score on a scale
  Readiness at baseline | 6.9 (3.5)
  Readiness immediately post intervention (day 1) | 7.7 (3.2)
  Readiness Post-intervention Day 30 | 7.1 (3.7)
  Importance at baseline | 7.7 (3.2)
  Importance immediately post intervention (day 1) | 7.5 (3.3)
  Importance Post-intervention Day 30 | 7.0 (3.6)
  Confidence at baseline | 6.9 (3.4)
  Confidence immediately post intervention (day 1) | 7.5 (3.5)
  Confidence Post-intervention Day 30 | 7.7 (3.3)

7. Primary Outcome: Participants Readiness to Change Alcohol Use
Description: The mean score of participants responses by self report. Participants were asked "If your provider felt it was a good idea, how ready are you to decrease your alcohol use?", "If your provider felt it was a good idea, how important is it for you to decrease your alcohol use?", and "If your provider felt it was a good idea, how confident are you that you can decrease your alcohol use?" Each question is scored on a 1-10 scale (1=not at all ready, 10=extremely ready). Total score range for each question is 1-10 with higher scores indicating better outcomes.
Time Frame: baseline, immediately post intervention (day 1) and Post-intervention Day 30
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 38
score on a scale
  Readiness at baseline | 6.4 (3.4)
  Readiness immediately post intervention (day 1) | 7.8 (3.4)
  Readiness Post-intervention Day 30 | 7.0 (3.7)
  Importance at baseline | 6.1 (3.8)
  Importance immediately post intervention (day 1) | 7.6 (3.4)
  Importance Post-intervention Day 30 | 6.83 (3.8)
  Confidence at baseline | 8.4 (2.5)
  Confidence immediately post intervention (day 1) | 8.9 (2.5)
  Confidence Post-intervention Day 30 | 8.7 (2.4)

8. Primary Outcome: Medication Use to Assess Acceptability
Description: The number of respondents who reported they (1) felt comfortable with the way medication information was presented, (2) understood the information given, (3) found the information helpful, (4) felt the amount of information was adequate, and (5) felt the information that they received was clear. Participants provided their responses to each question using a 5-point Likert scale (response options 1-5 with higher numbers indicating better acceptability). We will evaluate the number of participants who responded with a 4 or a 5.
Time Frame: Post-intervention Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 35
Participants
  Felt comfortable with the way medication information was presented | 23
  Understood the information given | 35
  Found the information helpful | 31
  Felt the amount of information was adequate | 32
  felt the information that they received was clear | 33

9. Primary Outcome: Information Regarding PEth to Assess Acceptability
Description: The number of respondents who reported that they (1) felt comfortable with the way PEth information was presented, (2) understood the information given, (3) found the information helpful, (4) felt the amount of information was adequate, and (5) felt the information that they received was clear. Participants provided their responses to each question using a 5-point Likert scale (response options 1-5 with higher numbers indicating better acceptability). We will evaluate the number of participants who responded with a 4 or a 5.
Time Frame: Post-intervention Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 35
Participants
  Felt comfortable with the way PEth information was presented | 25
  Understood the information given | 29
  Found the information helpful | 27
  Felt the amount of information was adequate | 6
  Felt the information that they received was clear | 30

10. Primary Outcome: General Feedback to Assess Acceptability
Description: The number of respondents who (1) felt they learned new things about their health risk from alcohol, (2) learned new things about their health risk from polypharmacy, (3) learned how medications and alcohol can act together, and (4) felt that having a pharmacist to talk with was helpful. Participants provided their responses to each question using a 5-point Likert scale (response options 1-5 with higher numbers indicating better acceptability). We will evaluate the number of participants who responded with a 4 or a 5.
Time Frame: Post-intervention Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Medications and Alcohol Use
Number analyzed (Participants) | 35
Participants
  Felt they learned new things about their health risk from alcohol | 19
  Learned new things about their health risk from polypharmacy | 29
  Learned how medications and alcohol can act together | 30
  Felt that having a pharmacist to talk with was helpful | 23

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | HIV Medications and Alcohol Use
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 1/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV Medications and Alcohol Use (N=38)
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Patient left study temporarily for health reasons prior to intervention activities, then returned to participate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT05560932/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT05560932/SAP_001.pdf
  • Informed Consent Form (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT05560932/ICF_002.pdf